CLINICAL TRIAL: NCT04637802
Title: Effectiveness of an mHealth Psychosocial Intervention to Prevent Transition From Acute to Chronic Postsurgical Pain in Adolescents
Brief Title: Digital Health Psychosocial Intervention for Adolescent Spine Surgery Preparation and Recovery
Acronym: SurgeryPal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Duke University (Other); University of Utah (Other); Vanderbilt University (Other); Johns Hopkins University (Other); Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Rabbitts, MBChB, Principal Investigator, Anesthesiologist, Seattle Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UH3HD102038 (NIH)
Record Dates: First submitted 2020-11-06; First posted 2020-11-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Juvenile; Scoliosis; Scoliosis Idiopathic; Scoliosis; Adolescence; Scoliosis;Congenital; Kyphosis; Spondylolisthesis
Keywords: Psychosocial Intervention; Spinal Fusion Surgery; Chronic Pain; Acute Pain; Adolescent; Randomized controlled trial
MeSH Terms: conditions — Scoliosis; Kyphosis; Spondylolisthesis; Chronic Pain; Acute Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized and double-blinded controlled trial of cognitive-behavioral intervention vs education at two phases (pre-operative and post-operative)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-operative and Post-operative Education intervention (Active Comparator): This arm receives access to Patient Education intervention in the pre- and post-operative phases.
  Interventions: Behavioral: Education
- Pre-operative CBT intervention (SurgeryPal), Post-operative Education intervention (Experimental): This arm receives access to CBT intervention in the pre-operative phase and Patient Education in the post-operative phase.
  Interventions: Behavioral: CBT (SurgeryPal); Behavioral: Education
- Pre-operative Education intervention, Post-operative CBT intervention (SurgeryPal) (Experimental): This arm receives access to Patient Education intervention during the pre-operative period and CBT intervention during the post-operative period.
  Interventions: Behavioral: CBT (SurgeryPal); Behavioral: Education
- Pre-operative and Post-operative CBT intervention (SurgeryPal) (Experimental): This arm receives access to CBT intervention during the pre-operative and post-operative period.
  Interventions: Behavioral: CBT (SurgeryPal)

INTERVENTIONS:
Behavioral: CBT (SurgeryPal) — The SurgeryPal intervention is a cognitive-behavioral program for youth undergoing major surgery. SurgeryPal is delivered in two 4-week phases: the pre-operative phase, and the post-operative phase. Each phase consists of 3 separate treatment modules for youth and parents, which teach cognitive and behavioral coping skills to target known psychosocial and behavioral risk factors (i.e. anxiety/distress and sleep disturbance) for poorer postsurgical outcomes, and provide training in pain self-management skills. Pre-operative modules include: 1) Preparing for surgery, 2) Coping with stress before surgery, and 3) Getting ready for the hospital. Postoperative modules include: 1) Coping at home after surgery, 2) Return to activities and school, and 3) Long-term recovery. Modules are self-guided and interactive, and focus on phases of preparation and recovery from surgery. The goal of the program is to reduce pain and enhance quality of life following surgery in youth.
  Arms: Pre-operative CBT intervention (SurgeryPal), Post-operative Education intervention; Pre-operative Education intervention, Post-operative CBT intervention (SurgeryPal); Pre-operative and Post-operative CBT intervention (SurgeryPal)
Behavioral: Education — The patient education website will serve as the active comparator. The purpose is to control for time, attention, and online usage. Youth and parents will be provided access to an education website containing information about pediatric surgery at the same time interval as the active intervention; however, there will be no exposure to cognitive and behavioral coping skills. Similar to the CBT condition, the presurgery period of Education will be administered for one month prior to surgery and the postsurgery period will be administered for one month after the post-discharge assessment.
  Arms: Pre-operative CBT intervention (SurgeryPal), Post-operative Education intervention; Pre-operative Education intervention, Post-operative CBT intervention (SurgeryPal); Pre-operative and Post-operative Education intervention

SUMMARY:
This is a randomized controlled trial to test effectiveness of the SurgeryPal intervention vs. education control to improve acute and chronic pain and health outcomes in youth undergoing major musculoskeletal surgery. Youth will be randomized on an individual level using a factorial design to SurgeryPal or Education during 2 phases of intervention: 1) pre-operative phase (4 week duration delivered over the 4 weeks leading up to surgery), and 2) post-operative phase (4 week duration following surgery). Thus there will be 4 treatment arms. Participants will undergo 4 assessments, independent of their treatment assignment: T1: Baseline (pre-randomization); T2: acute post-surgery outcomes (daily assessment of acute outcomes beginning day 1 through day 14 after hospital discharge from surgery); T3: Post-surgery follow-up (assessment of outcomes at 3-months post-surgery); T4: Final post-surgery follow-up (assessment of outcomes at 6-months post-surgery).

DETAILED DESCRIPTION:
Major musculoskeletal surgeries are associated with particularly high prevalence of both acute and chronic post-surgical pain (CPSP), with 80% of youth reporting intense acute pain after hospital discharge, and up to half reporting CPSP up to one year after spine surgery. Interventions to improve recovery and reduce pain after surgery have potential to interrupt a negative trajectory of suffering and disability associated with chronic pain. Our specific aims are: Primary: (1) Determine effectiveness of a pre-operative mHealth psychosocial intervention to improve acute pain outcomes in adolescents undergoing major musculoskeletal surgery, (2) Determine effectiveness of a post-operative mHealth psychosocial intervention to improve chronic pain outcomes at 3 months in adolescents undergoing major musculoskeletal surgery, (3) Determine the combined effects of pre- and post-operative psychosocial intervention on chronic pain outcomes. Secondary: (1) Determine effectiveness of pre-operative psychosocial intervention to reduce opioid use during the 14 days following hospital discharge, (2) Determine effectiveness of psychosocial intervention to improve health-related quality of life following surgery.

ELIGIBILITY:
Inclusion Criteria:

Teen

* 12 to 18 years old at the time of enrollment
* Undergoing scheduled spinal fusion surgery (eligible indications: juvenile/adolescent idiopathic scoliosis, congenital scoliosis, spondylolisthesis or kyphosis)

Parent/Caregiver

* Parent or legal guardian of child who meets study criteria

Exclusion Criteria:

Teen

* Does not speak or understand English
* Has severe learning disability, cognitive impairment or intellectual delay (i.e. unable to read at 5th grade level)
* Does not have access to a smart device (smartphone, iPad or tablet; Teens can borrow an iPad from the study team if one is available)
* Recent psychiatric admission (in the past 30 days)
* Severe systemic disease (neuromuscular scoliosis, cancer)
* On a regular treatment regimen for a severe chronic medical condition
* Prior major surgery (open surgery such as heart, lung, brain, abdominal surgery, or prior spine surgery)
* Diagnosed chronic musculoskeletal pain condition (e.g. complex regional pain syndrome, fibromyalgia, widespread musculoskeletal pain)

Parent/Caregiver

* Does not speak or understand English
* Does not have access to a smart device (smartphone, iPad or tablet)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 433 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Post-surgical pain intensity and interference | Up to 3 weeks post-surgery
  The Brief Pain Inventory (BPI) has 2 scales: pain intensity (4 items) and pain interference (7 items). Items are averaged to yield scale scores, ranging from 0 to 10, with higher scores indicating greater pain intensity or interference. The 24 hour (short) version of this measure will be completed via REDCap daily for 14 days post-hospital discharge (beginning on day 1 after hospital discharge, and ending up to 3-weeks post-surgery).
Chronic pain intensity and interference | 3 months post-surgery
  The Brief Pain Inventory (BPI) has 2 scales: pain intensity (4 items) and pain interference (7 items). Items are averaged to yield scale scores, ranging from 0 to 10, with higher scores indicating greater pain intensity or interference. The 24 hour (short) version of this measure will be completed via REDCap daily for 7 days at 3 months after the participant's surgery date.

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline, 3-months post-surgery, 6-months post-surgery
  The Pediatric Quality of Life Inventory (Peds-QL) 15-item short form assesses several domains of functioning, including physical, social, emotional, and academic functioning. The PedsQL is widely used and demonstrates good reliability for both the parent and child self-report measures. Scale scores range from 0 to 100. Higher scores indicate fewer difficulties (better) health-related quality of life. Subscales of physical and psychosocial health will be used in analyses.
Change in opioid use | Baseline, Up to 3 weeks post-surgery, 3-months post-surgery, 6-months post-surgery
  Youth will report medication use on the Brief Pain Inventory (BPI), including selecting medication name from a dropdown list (opioid, acetaminophen, anti-inflammatory, other). Number of days of opioid use will be used in analyses.
Change in opioid misuse | Baseline, 3-months post-surgery, 6-months post-surgery
  The American Psychiatric Association (APA) Adapted National Institute for Drug Abuse (NIDA) Modified Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) Level 2 Tool (Teen Report) recommended by the National Institute on Drug Abuse for substance use screening in adolescents, will be used to assess alcohol, smoking, substance, and opioid use. Additional questions on reasons for misuse (e.g. to treat pain, to get high, etc.) and source of opioids (e.g. prescription, from a friend or relative) will be collected using the corresponding questions and response options used in the National Survey on Drug Use and Health.
Change in psychosocial distress | Baseline, 3-months post-surgery, 6-months post-surgery
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Emotional Distress Scales include an 8-item scale of anxiety that assesses fear (e.g., fearfulness), anxious misery (e.g., worry) and hyperarousal (e.g., nervousness) and 8-item scale of depressive symptoms that evaluates negative mood, view of self and social cognitions. Response options range from 1 (Never) to 5 (Almost Always). Raw scores for anxiety and depression are obtained by summing the corresponding items' response values, and range from 8 to 40 with higher scores indicating higher distress.
Change in mental health | Baseline, 3-months post-surgery, 6-months post-surgery
  Parents and teens will self-report on the Patient Health Questionnaire-4, a 4 item screening measure of general anxiety and depressive symptoms. Response options range from 0 (Not at all) to 3 (Nearly Every Day). Total scores are calculated by summing items, for a total score ranging from 0 to 12, with higher scores indicating greater anxiety and depressive symptoms.
Change in sleep quality | Baseline, 3-months post-surgery, 6-months post-surgery
  The Adolescent Sleep Wake Scale 10-item version (Teen Report) is a 10-item measure assesses self-reported sleep quality. Scale scores range from 1 to 6 with higher scores indicating better sleep quality. Four additional items assess sleep duration on weekdays and weekends.
Change in pain catastrophizing | Baseline, 3-months post-surgery
  The Pain Catastrophizing Scale - Child Version and Parent Version is a Self-report 13 item measures that assess child pain catastrophizing and parent's catastrophizing about child's pain, respectively. Total scores range from 0 to 52 with higher scores indicating greater pain catastrophizing.
Global pain severity | Up to 3 weeks post-surgery, 3-months post-surgery, 6-months post-surgery
  The Patient Global Impression of Severity Scale (PGIS), Teen Report is a 1-item measure that assesses adolescent's self-reported global impression of pain severity. Response options range from 0 (none) to 3 (severe) with higher scores indicating higher pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rabbitts, MD, Principal Investigator — Seattle Children's Hospital; Tonya Palermo, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A releasable database for underlying primary data for publications will be made broadly available on the NIH HEAL Initiative central data repository. The database will be produced and will be completely de-identified in accordance with the definitions provided in the Health Insurance Portability and Accountability Act (HIPAA). The DCC will also prepare a data dictionary that provides a concise definition of every data element included in the database. In accordance with policies of the NIH, the DCC will send the releasable database to the entity determined by the NIH or specific institute to be the repository for data created under the HEAL initiative. The DCC is able to produce a relational database export, or use SAS or SPSS data sets. The DCC will accompany the database with full documentation so that individual investigators will be able to effectively use the data.
Time Frame: After last subject enrollment and all follow up procedures have been completed, the HEAL Pain Management Effectiveness Research Network Data Coordinating Center (DCC) at the University of Utah will prepare a final study database for the trial, which will then be used for statistical analyses and publication of findings from the trial. The policies for release of this database are in accordance with the HEAL Data Sharing policy as determined by the NIH. Our preliminary plan is to release the underlying primary database at the time of publication of the primary manuscript. The primary publication from the dataset will be made publicly available immediately without any embargo period through the Creative Commons Generic License in accordance with the HEAL Public Access guidance. Additional secondary publications will be deposited electronically within 4 weeks of acceptance into PubMed Central.
Access Criteria: Access to the releasable database housed in the NIH-assigned repository will be in accordance with procedures and regulations of the NIH or specific institute. The DCC will not provide any support for investigators using the releasable database.

REFERENCES:
- [Derived] Rabbitts JA, Zhou C, de la Vega R, Aalfs H, Murray CB, Palermo TM. A digital health peri-operative cognitive-behavioral intervention to prevent transition from acute to chronic postsurgical pain in adolescents undergoing spinal fusion (SurgeryPalTM): study protocol for a multisite randomized controlled trial. Trials. 2021 Jul 30;22(1):506. doi: 10.1186/s13063-021-05421-3. PMID 34330321